CLINICAL TRIAL: NCT05985486
Title: The Impact of Weight Loss on Alzheimer's Disease Risk in Adults With Down Syndrome
Brief Title: Brain Outcomes With Lifestyle Change in Down Syndrome
Acronym: BOLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Study 150542
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Down Syndrome; Alzheimer Disease; Obesity
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease; Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Loss (Experimental): * Follow a reduced calorie diet daily for 12 months.
  * Attend monthly behavioral counseling/education
  Interventions: Behavioral: Diet; Behavioral: Health Education
- General Health Education Control (Active Comparator): - Attend monthly health education sessions about general health.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Diet — A reduced calorie diet which uses frozen meals purchased at the store and focuses on increasing fruits and vegetables associated with brain health.
  Arms: Weight Loss
Behavioral: Health Education — Monthly health education sessions delivered remotely.

SUMMARY:
The goal of this study is to determine if weight loss or changes in dietary intake can help prevent of delay adults with Down syndrome from developing Alzheimer's Disease

Adults with Down syndrome without dementia will be randomized to either a weight loss group or a general health education control group. The weight loss group will be asked to follow a reduced energy diet, attend monthly education sessions delivered remotely and self-monitor diet and body weight using commercially available web-based applications. The control group will be asked to attend remotely delivered monthly education sessions on general health education topics.

All participants will come to the University of Kansas Medical Center, 3 times across 12 months for a blood draw, cognitive testing, a MRI, assessment of height and weight, and assessment of diet intake.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome
* BMI of 25 to 50 kg/m2
* Ability to communicate through spoken language.
* Ability to come to the University of Kansas Medical Center 3 times across 1 year for outcomes testing
* Living at home with a parent/guardian, or in a supported living environment with a caregiver who assists with food shopping, meal planning, and meal preparation and agrees to serve as a study partner including providing transportation to our facilities for study assessments.

Exclusion Criteria:

* Diagnosis of dementia
* Insulin dependent diabetes
* Participation in a weight management program involving diet or physical activity in the past 6 mos.
* Dairy allergy
* Serious medical risk (e.g., cancer, recent heart attack, stroke, pregnancy, angioplasty)
* Unwilling to be randomized
* Contraindications for MRI, including metal implants or devices incompatible with MRI such as pacemakers, claustrophobia, and inability to lay in a supine position
* Use of GLP-1 medications
* Use of anti-amyloid medications

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Amyloid beta 42:40 ratio | Baseline, 6, 12 months
  Examines the amount of amyloid beta in a person's brain, measured by a blood draw.
Neurofilament light | Baseline, 6, 12 months
  Examines the amount of Neurofilament light in a person's brain, measured by a blood draw.
Weight | Baseline, 6, 12 months
  Examines how much a person weights, measured by standing on a scale.

SECONDARY OUTCOMES:
Dietary Intake | Baseline, 6, 12 months
  Examines what someone is eating, measured by writing down what a person eats over 3 days.
Skin carotenoid content | Baseline, 6, 12 months
  Examines how many vegetables a person eats, measured by a finger scan using the Veggie Meter.
Plasma Phosphorylated Tau | Baseline, 6, 12 months
  Examines the amount of Tau in a person's brain, collected by a blood draw.
Glial Fibrillary Acidic Protein | Baseline, 6, 12 months
  Examines the amount of Glial Fibrillary Acidic Protein in a person's brain, collected by a blood draw.
Brian Volume | Baseline, 12 months
  Examines how much white and grey matter a person has in their brain, measured by MRI
Brain antioxidants | Baseline, 12 months
  Examines the amount of GHS and vitamin C a person has in their brain. Measured by MRI
The modified Cued Recall Test | Baseline, 6, 12 months
  Measures cognitive function. Twelve items are presented for learning, 4 at a time, with each item accompanied by a unique category cue. The testing phase consists of 3 trials. Each trial begins with free recall of the test items; following free recall, a category cue is provided for those items not spontaneously recalled.
The Modified Cats and Dogs Task | Baseline, 6, 12 months
  Measures executive function. The task measures the ability to inhibit a natural response (naming the pictures of a dog, as "dog") and to replace it with an incongruent one (naming the pictures of a dog as "cat").
Down Syndrome Mental Status Examination | Baseline, 6, 12 months
  Provides an omnibus measure of neuropsychological functioning, assessing recall of personal information, orientation, immediate and delayed memory, language, visuospatial function and praxis.

OTHER OUTCOMES:
Height | Baseline, 6, 12 months
  Examines how tall a person is, measured on a stadiometer
Waist circumference | Baseline, 6, 12 months
  Examines the distance around the smallest part of a person's torso, measured with a measuring tape
Attendance at education sessions | Across 12 months
  Examines how often individuals attendance the monthly education sessions. Obtained from interventionist records and expressed as the percentage of possible sessions attended.
Compliance with self-monitoring of diet | Across 12 months
  Assessed as the percentage of days a person tracked what they ate across the study.
Physical Activity | Baseline, 6, 12 months
  Examines Daily minutes of light, moderate, and vigorous physical activity as well as sedentary time using an ActiGraph tri-axial accelerometer worn on a wrist for 7 days.
Structured interviews | 12 months
  A 20% random sample of participants and study partners from each intervention arm will complete a 30 minute interview to gather information that might be useful for improving the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No